CLINICAL TRIAL: NCT06270121
Title: Development of an Integrated Contactless Healthcare Service Platform Based on Intelligent IoT for the Successful Aging of the Elderly
Brief Title: Development of a Healthcare Service Platform for Successful Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunmi Song (Other)
Responsible Party: Sponsor-Investigator, Sunmi Song, Research Professor, Korea University
Organization: Korea University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: R2111483
Record Dates: First submitted 2023-11-01; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Depression in Old Age; Chronic Pain; Sleep Disorder Insomnia Chronic
Keywords: geriatric depression; digital mental health phenotyping; community based hybrid digital senior care service; digital healthcare monitoring platform for elderly; chronic pain; sleep disorders
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Control group was informed that they participated in the study with a repeated measure survey about digital healthcare for elderly without detailed descriptions on the living-lab intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living-lab digital intervention group (Experimental): Digital devices (wearable and motion sensor) and mobile application will be utilized to monitor mental and physical health status and provide daily individualized health status information to an older adult user and their community and family caregivers. The older adult users are also asked to participate in pre-mid-post surveys to evaluate health, usability, effectiveness, and safety of the developed platform service.
  Interventions: Behavioral: Living-lab digital intervention group
- Control group (No Intervention): The participated in the control group are asked to participate in pre-mid-post surveys to evaluate health status.

INTERVENTIONS:
Behavioral: Living-lab digital intervention group — Older adults will receive individualized daily health feedback via the mobile applications, which will be shared with caregivers. They will also receive support for health emergency by the platform sending automatic emergency push alarm to community and family caregivers.
  Arms: Living-lab digital intervention group

SUMMARY:
The goal of this living-lab clinical trial is to test the effectiveness of digital health monitoring and feedback platform for community dwelling older adults. The main questions it aims to answer are:

* Identify digital sensing variables that are predictive of mental and physical health declines and health emergencies of older adults
* Develop digital health monitoring service to inform individualized daily health status of older adults users
* Develop ICT network to share the daily health status and emergency signals with community based healthcare service providers and family caregivers if an older adult user approves of them to receive their health information.

Participants will be asked to participate in a living lab using a wearable sensor, motion sensor, and smartphone applications for 6 weeks and also take part in pre-mid-post surveys to evaluate the usability, accuracy, and effectiveness of the digital healthcare service platform to improve health managements and connections with community and family caregivers.

If there is a comparison group: Researchers will compare age and gender matched control group to see if health status of the living-lab group is better than the control group.

DETAILED DESCRIPTION:
The purpose of the living-lab clinical trials is to develop contactless digital health monitoring system and individually customizable health status feedback contents in order to improve self-care capacity and mental health of older adults who live alone. Also, the current trials aim to evaluate effectiveness and usability of the overall developed monitoring platform. The effectiveness evaluation will investigate whether the platform can be effective at detecting levels of health decline or improvements and connecting in-person healthcare services. The usability tests will focus on user-centeredness, efficiency, and usability for older adults and their community healthcare provider.

To accomplish the purposes, the platform was developed based on needs assessments and observations of living environments of community dwelling older adults using surveys and interviews. Community healthcare providers also participated interview on their needs as a caregiver and working conditions that need to be considered to develop applications and website for community caregivers.

The developed platform will be tested by younger adults for a pilot test and be tested by older adult users and their matched controls for the main clinical trials. The older adults participants will be recruited via postings and study information sessions at the community senior welfare center in Seoul, South Korea. Interested older adults and community healthcare service providers will be invited to participation in the trials. After recruiting the living lab older adults, age and gender matched control older adults will be recruited. Older adult participants will be those who are over 65 years old and do not have cognitive and sensory disorders (e.g., deafness or dementia) that may inhibit participation in the trials.

The living lab will be conducted for 6 weeks, starting with a 1-week adaptation period. Older adults will be asked to open the smartphone application in the morning; the application would automatically link them to a chatbot asking how they are doing and 2 questions on daily depressive symptoms.

After using the chatbot, the participants will be able to see their daily health status information for stress (via high frequency measure (HF) of heart rate variability (HRV)), sleep (via total sleep time and sleep fragmentation), and physical activity (via steps) on the previous day, compared to their own average during the first week of the living lab.

Their voice records and daily health status will be sent to their matched community caregiver via a study website. A manager at the senior welfare center will be able to monitor any health emergency by participated older adults via the study website.

During the living lab period, the older adult participants will be asked to wear a smartwatch continuously except while the battery is being charged. For the effectiveness and usability evaluations, both living lab and control participants will be invited to surveys before, during, and after the 6 week periods. Community caregivers and managers will evaluate the effectiveness and usability via a survey and interview after the 6 week living lab period.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling older adults who are 65 years old and older

Exclusion Criteria:

* Older adults with cognitive, sensory, and functional problems that may hinder them from participating surveys.
* Older adults with iOS mobile device that would not allow them to use the developed mobile application.
* Older adults in nursing home or who are hospitalized because this platform is designed to support independent living of an older adults in their home.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Daily assessments across 6 weeks
  PHQ-9 items will be used to assess daily depressive symptoms using a chatbot, the total score ranged from 0 to 27, higher score representing more severe depressive status.
Sleep fragmentation index | Daily assessments across 6 weeks
  Number of awakening divided by total sleep time in percentage, ranged from 0 to 100, higher score indicating more fragmented sleep.
Daily steps | Daily assessments across 6 weeks
  Number of steps per day, which can be ranged from 0 to infinite. Higher numbers of steps indicate more physical activity for the day.
Intensity of physical activity | Daily assessments across 6 weeks
  Minutes of light, moderate, and intense physical activity, which can be ranged from 0 to 1440 minutes. More active minutes at each of the three intensity levels presents more physical activities.
Heart rate variability | Daily assessments across 6 weeks
  Daily assessments of heart rate variability

SECONDARY OUTCOMES:
Geriatic depression | Before and after the 6 week living lab periods
  Geriatric depression scale score ranges from 0-15 with higher scores indicating more severe depressive symptoms.
SF-12 Quality of life | Before and after the 6 week living lab periods
  Short Form survey-12 (SF-12) measures levels of the health related quality of life, which ranges from 0 to 100 with higher scores presenting better quality of life.
Pain related functional limitations | Before and after the 6 week living lab periods
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), which ranged from 0 to 90 with higher scores indicating worse pain related functional limitations in one's daily living.
Chronic pain | Before and after the 6 week living lab periods
  Brief Pain Inventory (BPI) score ranges from 1 to 10 with higher score indicating more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Junesun Kim, PhD, Principal Investigator — Korea University
Locations (1):
- Korea University, Seoul, South Korea

REFERENCES:
- [Derived] Song S, Seo Y, Hwang S, Kim HY, Kim J. Digital Phenotyping of Geriatric Depression Using a Community-Based Digital Mental Health Monitoring Platform for Socially Vulnerable Older Adults and Their Community Caregivers: 6-Week Living Lab Single-Arm Pilot Study. JMIR Mhealth Uhealth. 2024 Jun 17;12:e55842. doi: 10.2196/55842. PMID 38885033